CLINICAL TRIAL: NCT01579942
Title: Potential Use Of Brain Network Activation Analysis Using Evoked Response Potentials to Diagnose Major Depression and Assess Response to Antidepressant Treatment
Brief Title: Potential Use Of Brain Network Activation Analysis to Diagnose Major Depression
Status: Terminated | Type: Observational
Why Stopped: The study was ultimately not funded by the sponsor. No subjects were enrolled.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ElMindA Ltd (Industry)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2011P000200
Record Dates: First submitted 2012-04-11; First posted 2012-04-18 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Major Depressive Disorder
Keywords: EEG; Biomarker; Major Depressive Disorder; Healthy Control
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Major Depressive Disorder: Patients who have Major Depressive Disorder and are taking a Selective Serotonin Re-uptake Inhibitor (SSRI) as part of another study at our clinic.
- Healthy Controls: Patient with no history of significant mental health problems.

SUMMARY:
The investigators are doing this study to find out if they can use electroencephalographic (EEG) recordings, which measure brain waves, to predict response to antidepressant treatments, as well as to distinguish patients who have depression from those who do not. In particular the investigators want to test the usefulness of a new type of analysis of EEG recordings called brain network activation or BNA. BNA allows to identify patterns of activation in brain networks and to track their changes over time.

ELIGIBILITY:
For Patients with Major Depressive Disorder

Inclusion Criteria:

* • Male and female outpatients, aged 18-55 years

  * Subjects meeting full criteria for the diagnosis of current Major Depressive Disorder (MDD) without psychotic features, as determined by clinical evaluation and Mood Module of structured diagnostic interview (SCID), completed by the study clinician.
  * HAM-D17 score of 14 or higher
  * Able to provide informed consent
  * Right handed, normal (corrected) vision and normal hearing

Exclusion Criteria:

* • Other primary diagnoses including major depressive disorder with psychotic features, bipolar disorder, schizoaffective disorder, schizophrenia, dementia, attention deficit hyperactivity disorder (ADHD).

  * Substance use disorder (abuse or dependence with active use within the last 6 months).
  * Significant sensory deficits such as deafness or blindness.
  * Severe or unstable medical illness, including history of closed head injury resulting in loss of consciousness, seizure disorder; history of neurological disorders.
  * Pregnant or nursing females who are not using an accepted method of contraception (birth control pill, IUD, combination of barrier methods)
  * Clinically significant abnormal laboratory values or electrocardiogram For Healthy Controls

Inclusion Criteria:

* Males and females, aged 18-55 years
* Subjects who do not meet full criteria for any of the major psychiatric diagnosis including MDD, bipolar disorder, schizophrenia, substance abuse/dependence, attention deficit hyperactivity disorder (ADHD), as determined by clinical evaluation and structured diagnostic interview, completed by the study clinician.
* Right handed, normal (corrected) vision and normal hearing

Exclusion Criteria:

* Any current primary psychiatric, or medical condition determined to be clinically significant.
* Current use of psychotropics or any medication with clinically significant central nervous system effects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For Patients with Major Depressive Disorder
  • Subjects meeting full criteria for the diagnosis of current Major Depressive Disorder (MDD) without psychotic features, as determined by clinical evaluation and Mood Module of structured diagnostic interview (SCID), completed by the study clinician.
  For Healthy controls
  * Males and females, aged 18-55 years
  * Subjects who do not meet full criteria for any of the major psychiatric diagnosis including MDD, bipolar disorder, schizophrenia, substance abuse/dependence, as determined by clinical evaluation and structured diagnostic interview, completed by the study clinician.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2012-04

PRIMARY OUTCOMES:
Brain Network Analysis group patterns | 8 weeks
  The investogators will make a comparison of Functional networks of brain activity (BNA™) in subjects with MDD and healthy individuals measured using analysis of EEG Event Related Potential (ERP) data [ Time Frame: Baseline, 1 week after the first dose of antidepressant treatment, end of the treatment phase].

SECONDARY OUTCOMES:
Identify possible predictors of treatment response | 8 weeks
  The investigators will examine the agreement between clinical diagnoses and the change of Brain Network Activation (BNA™)Scores in MDD subjects and healthy controls.
  Subjects will undergo clinical diagnostic interviews and a comprehensive neuropsychological and cognitive assessment, and then complete 1 EEG scan of approximately 1 hour. The results of the BNA will be compared to the results of the clinical diagnostic interviews and tests.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Cusin, MD, Principal Investigator — Massachusetts General Hospital; Ottavio Vitolo, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program, Boston, Massachusetts, United States